CLINICAL TRIAL: NCT03816332
Title: Immune Checkpoint Blockade for Kidney Transplant Recipients With Selected Unresectable or Metastatic Cancers
Brief Title: Tacrolimus, Nivolumab, and Ipilimumab in Treating Kidney Transplant Recipients With Selected Unresectable or Metastatic Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-00239; NCI-2019-00239 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ETCTN10214; 10214 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10214 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2019-01-24; First posted 2019-01-25 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage III Cutaneous Merkel Cell Carcinoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Merkel Cell Carcinoma AJCC v8; Metastatic Basal Cell Carcinoma; Metastatic Melanoma; Metastatic Merkel Cell Carcinoma; Metastatic Skin Squamous Cell Carcinoma; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage III Cutaneous Merkel Cell Carcinoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Cutaneous Merkel Cell Carcinoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Merkel Cell Carcinoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Merkel Cell Carcinoma AJCC v8; Unresectable Basal Cell Carcinoma; Unresectable Melanoma; Unresectable Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Melanoma; Carcinoma, Merkel Cell | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; Prednisone; deltacortene; prednylidene; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tacrolimus, prednisone, nivolumab, ipilimumab) (Experimental): Patients receive tacrolimus PO BID and prednisone PO QD. Within 28 days, patients then receive nivolumab IV over 30 minutes on day 1. Cycles repeat every 4 weeks for up to 24 cycles (96 weeks) in the absence of disease progression or unacceptable toxicity.
  Patients who experience PD or patients who have experienced allograft loss at 16 weeks receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1. Patients also receive tacrolimus PO BID and prednisone PO QD. Cycles repeat every 3 weeks for 4 cycles (12 weeks) in the absence of disease progression or unacceptable toxicity. Starting 6 weeks later, patients receive nivolumab IV over 30 minutes every 4 weeks for up to 21 cycles (84 weeks) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Drug: Prednisone; Drug: Tacrolimus

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Drug: Tacrolimus — Given PO
  Other Names: FK 506; FK-506; FK506; Fujimycin; Hecoria; Prograf; Protopic; Tacforius

SUMMARY:
This phase I trial studies how well tacrolimus, nivolumab, and ipilimumab work in treating kidney transplant recipients with cancer that cannot be removed by surgery (unresectable) or has spread to other places in the body (metastatic). Tacrolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving tacrolimus, nivolumab, and ipilimumab may work better in treating kidney transplant recipients with cancer compared to chemotherapy, surgery, radiation therapy, or targeted therapies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the percent of kidney transplant recipients with selected advanced cancers for whom standard therapies would be insufficient who, 16 weeks after administration of prednisone, tacrolimus, and nivolumab, experience complete response (CR), partial response (PR), or stable disease (SD) without allograft loss.

SECONDARY OBJECTIVES:

I. To estimate the objective response rate (ORR), rate of allograft loss, and durations of progression-free survival (PFS) and overall survival (OS) in the study population.

II. To estimate the ORR and rate of allograft loss in patients who experience progressive disease (PD) after administration of nivolumab and 1) receive ipilimumab and nivolumab, or 2) decrease or discontinue immunosuppression.

EXPLORATORY OBJECTIVES:

I. To characterize correlates of the host immune response, possibly including, but not limited to:

Ia. Histopathological characteristics of allograft rejection/loss. Ib. Immunological changes in the tumor microenvironment (e.g., changes in T-cell subset populations or expression of immune checkpoint molecules) in paired biopsies obtained pre-treatment and on-treatment.

Ic. Changes in donor-derived cell-free deoxyribonucleic acid (DNA) (dd-cfDNA) as a marker for allograft rejection.

Id. Characteristics of anti-programmed death-1 (PD-1)-associated immune-mediated adverse reactions (IMAR) in this patient population treated with immunosuppression.

OUTLINE:

Patients receive tacrolimus orally (PO) twice daily (BID) and prednisone PO once daily (QD). Within 28 days, patients then receive nivolumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 4 weeks for up to 24 cycles (96 weeks) in the absence of disease progression or unacceptable toxicity.

Patients who experience progressive disease (PD) or patients who have experienced allograft loss at 16 weeks receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1. Patients also receive tacrolimus PO BID and prednisone PO QD. Cycles repeat every 3 weeks for 4 cycles (12 weeks) in the absence of disease progression or unacceptable toxicity. Starting 6 weeks later, patients receive nivolumab IV over 30 minutes every 4 weeks for up to 21 cycles (84 weeks) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 90 days, every 8 weeks for year 1, every 12 weeks for year 2, every 16 weeks for year 3, then every 24 weeks for year 4. Patients with PD are followed up every 12 weeks for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be kidney transplant recipients with a functioning allograft who do not currently require dialysis
* Patients must have histologically or cytologically confirmed melanoma, basal cell carcinoma, Merkel cell carcinoma, cutaneous squamous cell carcinoma, or microsatellite instability (MSI)-high cancers for which standard non-immunological medical, surgical, or radiation therapy would be insufficient (i.e., patients who are not surgical candidates). This trial is not intended to provide therapy as a neoadjuvant approach
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, i.e., at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm by chest x-ray or as >= 10 mm with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam is preferred, but not required. Patients with evaluable disease but no target lesions (e.g., evaluable bone metastases) may be included after discussion with the principal investigator (PI)
* Patients must have documentation, in consultation with the PI, that they received, refused, or were ineligible for the following non-immunologic therapies:

  * For patients with:

    * BRAF-mutant melanoma: prior therapies include BRAF/MEK inhibitors
    * Merkel cell carcinoma: prior therapies include platinum + VP-16
    * Basal cell carcinoma: prior therapies include Hedgehog pathway inhibitors
    * Cutaneous squamous cell carcinoma: prior therapies include cetuximab
    * MSI colorectal carcinoma: prior therapies include: leucovorin calcium, 5-fluorouracil and oxaliplatin (FOLFOX)
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Serum creatinine =< 3 x ULN

  * Note: patients with creatinine levels above 3 x ULN may be eligible after consultation with the study PI
* The effects of nivolumab and ipilimumab on the developing human fetus are unknown. For this reason, and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (e.g., hormonal or barrier methods of birth control, or abstinence) prior to study entry, for the duration of study participation, and for 31 weeks after the last dose of nivolumab or ipilimumab. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of beta-human chorionic gonadotropin [B-HCG]) during the screening period. Follow-up evaluations will include interval sexual/menstrual histories as needed. Men who receive nivolumab or ipilimumab and are sexually active with WOCBP must use a contraceptive method with a failure rate of < 1% per year for the duration of the study and for a period of 7 months after the last dose of nivolumab or ipilimumab. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) should inform the treating physician immediately. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. Women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL to be considered postmenopausal
* Human immunodeficiency virus (HIV)-infected patients will be eligible for this trial if they are on effective antiretroviral regimens utilizing non-CYP-interactive agents and have an undetectable viral load. If there is evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy, if indicated. If there is history of hepatitis C virus (HCV) infection, the patient must have been treated and have undetectable HCV viral load
* Patients must be able to understand and be willing to sign a written informed consent document

Exclusion Criteria:

* Patients must not have received a liver, lung, heart, or pancreas transplant; or allogeneic stem cell transplant; or any kind of bone marrow transplant
* Patients must not be unwilling or unable to undergo dialysis
* Patients must not have prior evidence of human leukocyte antigen (HLA) or non-HLA donor-specific antibodies (DSA). Patients with detectable DSA but negative dd-cfDNA may be eligible after consultation with the study PI
* Patients must not have a history of antibody- or cell-mediated allograft rejection within 3 months of study entry
* Patients must not have had chemotherapy or radiotherapy within 4 weeks of study entry or those who have not recovered from adverse events (AEs) due to agents administered more than 4 weeks earlier
* Patients must not have had prior treatment for their current cancer with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Patients must not be receiving any other investigational agents
* Patients must not have known central nervous system (CNS) metastases or leptomeningeal metastases because of poor prognosis and concerns regarding progressive neurologic dysfunction that would confound the evaluation of neurologic and other AEs. Patients with brain metastases are permitted to enroll if metastases have been treated and there is no MRI evidence of progression for 4 weeks after treatment is complete and no evidence of progression within 28 days prior to study entry
* Patients must not have a history of severe hypersensitivity reaction to any monoclonal antibody
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to other agents used in study
* Patients must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because nivolumab and ipilimumab have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated with nivolumab or ipilimumab. These potential risks may also apply to other agents used in this study
* Patients must not have active autoimmune disease, or history of autoimmune disease that might recur, which may affect vital organ function, and will only be eligible after consultation with the study PI

  * This includes but is not limited to:

    * Immune-related neurologic disease,
    * Multiple sclerosis,
    * Autoimmune (demyelinating) neuropathy,
    * Guillain-Barre (GB) syndrome,
    * Myasthenia gravis,
    * Systemic autoimmune diseases such as systemic lupus erythematosus (SLE),
    * Connective tissue diseases,
    * Scleroderma,
    * Inflammatory bowel disease (IBD; e.g., ulcerative colitis or Crohn's disease),
    * Rheumatoid arthritis, and
    * Sjogren's syndrome
* Patients must not have had evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2026-09-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Evan J Lipson, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (7):
- United States (7):
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Schenk KM, Deutsch JS, Chandra S, Davar D, Eroglu Z, Khushalani NI, Luke JJ, Ott PA, Sosman JA, Aggarwal V, Schollenberger MD, Sharfman WH, Bibee KP, Scott JF, Loss MJ, Wang H, Qi H, Sharon E, Streicher H, Chen HX, Woodward RN, Bagnasco SM, Taube JM, Topalian SL, Brennan DC, Lipson EJ. Nivolumab + Tacrolimus + Prednisone +/- Ipilimumab for Kidney Transplant Recipients With Advanced Cutaneous Cancers. J Clin Oncol. 2024 Mar 20;42(9):1011-1020. doi: 10.1200/JCO.23.01497. Epub 2024 Jan 22. PMID 38252910
- [Derived] Bonilla M, Gudsoorkar P, Wanchoo R, Herrmann SM, Jhaveri KD. Onconephrology 2022: An Update. Kidney360. 2023 Feb 1;4(2):258-271. doi: 10.34067/KID.0001582022. Epub 2022 Dec 9. PMID 36821617
- [Derived] Trager MH, Coley SM, Dube G, Khan S, Ingham M, Samie FH, Geskin LJ, McDonnell D, Brouder D, Saenger Y, Carvajal R. Combination checkpoint blockade for metastatic cutaneous malignancies in kidney transplant recipients. J Immunother Cancer. 2020 Jun;8(1):e000908. doi: 10.1136/jitc-2020-000908. PMID 32503950

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Patients received low-dose tacrolimus (serum trough goal 2-5 ng/mL), prednisone 5mg by mouth once a day, and nivolumab 480mg by infusion every 4 weeks for up to 96 weeks in the absence of disease progression or unacceptable toxicity.
  Patients who experienced disease progression by the 16-week time point, could receive tacrolimus, prednisone, nivolumab 3 mg/kg IV + ipilimumab 1 mg/kg by infusion every 3 weeks for 4 doses followed by maintenance nivolumab 480mg by infusion every 4 weeks for up to 96 weeks in the absence of disease progression or unacceptable toxicity.
Period: Nivolumab, Tacrolimus, and Prednisone
Arm/Group | Treatment
Started | 12
Completed | 8
Not Completed | 4
Not completed — Did not receive Nivolumab | 2
Not completed — Death | 2
Period: Nivolumab, Ipilimumab, Tacrolimus, Pred
Arm/Group | Treatment
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Tacrolimus, Prednisone, Nivolumab, Ipilimumab): Patients received low-dose tacrolimus (serum trough goal 2-5 ng/mL), prednisone 5mg by mouth once a day, and nivolumab 480mg by infusion every 4 weeks for up to 96 weeks in the absence of disease progression or unacceptable toxicity.
  Patients who experienced disease progression by the 16-week time point, could receive tacrolimus, prednisone, nivolumab 3 mg/kg IV + ipilimumab 1 mg/kg by infusion every 3 weeks for 4 doses followed by maintenance nivolumab 480mg by infusion every 4 weeks for up to 96 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (Tacrolimus, Prednisone, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 69 [44 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 12
Height [Median (Full Range); unit: centimeter (cm)] | 168.4 [145.5 to 189.0]
Weight [Median (Full Range); unit: kilogram (kg)] | 68.3 [46.4 to 104.7]
BSA [Median (Full Range); unit: meters squared (m^2)] | 1.74 [1.39 to 2.34]

OUTCOME MEASURES:

1. Primary Outcome: Number (and Percentage) of Outcome Responses After Receiving Nivolumab, Tacrolimus, and Prednisone
Description: Percentage of kidney transplant recipients who experienced complete response (CR), partial response (PR) or stable disease (SD) without allograft loss.
Time Frame: At 16 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Nivolumab, Tacrolimus, and Prednisone: Patients received low-dose tacrolimus (serum trough goal 2-5 ng/mL), prednisone 5 mg by mouth once a day, and nivolumab 480 mg by infusion over 30 minutes on day 1. Cycles repeated every 4 weeks for up to 24 cycles (96 weeks) in the absence of disease progression or unacceptable toxicity.
Arm/Group | Nivolumab, Tacrolimus, and Prednisone
Number analyzed (Participants) | 8
Participants
  Complete response (CR), partial response (PR) or stable disease (SD) without allograft loss | 0
  Progressive Disease (PD) without allograft loss | 8

2. Secondary Outcome: Objective Response (CR or PR) Rate (ORR) After Receiving Nivolumab, Tacrolimus, and Prednisone
Description: Number (and percentage) of patients with a complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria after receiving at least one dose of nivolumab.
Time Frame: Up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Tacrolimus, and Prednisone
Number analyzed (Participants) | 8
Participants
  Complete response (CR) or Partial Response (PR) | 0
  Progressive Disease (PD) | 8

3. Secondary Outcome: Rate of Allograft Loss After Receiving Nivolumab, Tacrolimus, and Prednisone
Description: Number of subjects who experienced allograft loss after receiving at least one dose of nivolumab.
Time Frame: Up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Tacrolimus, and Prednisone
Number analyzed (Participants) | 8
Participants
  Experienced allograft loss | 0
  Did not experience allograft loss | 8

4. Secondary Outcome: Duration of Progression-free Survival After Receiving Nivolumab, Tacrolimus, and Prednisone
Description: From the first dose of nivolumab to the date of the first documented tumor progression or death due to any cause, whichever occurs first.
Time Frame: Up to 4 months
Measure: Mean (Full Range); unit: days
Arm/Group | Nivolumab, Tacrolimus, and Prednisone
Number analyzed (Participants) | 8
days | 59 [54 to 70]

5. Secondary Outcome: Duration of Overall Survival After Receiving Nivolumab, Tacrolimus, and Prednisone
Description: The time from the participant's first dose of nivolumab to the date of death from any cause.
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Nivolumab, Tacrolimus, and Prednisone
Number analyzed (Participants) | 8
months | 9.1 [1.9 to 37.0]

6. Secondary Outcome: Overall Response Rate (ORR) in Patients After Receiving Ipilimumab, Nivolumab, Tacrolimus, and Prednisone
Description: The number of participants with a CR or PR response after receiving ipilimumab, nivolumab, tacrolimus, and prednisone.
Time Frame: Up to 3 years
Population: Two participants who completed the initial treatment period did not start the second, optional treatment period due to disease progression or death.
Measure: Count of Participants; unit: Participants
Groups:
- Ipilimumab, Nivolumab, Tacrolimus, and Prednisone: Patients received low-dose tacrolimus (serum trough goal 2-5 ng/mL), prednisone 5 mg every day, nivolumab 3 mg/kg by infusion and ipilimumab 1 mg/kg by infusion every 3 weeks for 4 doses followed by maintenance nivolumab 480mg by infusion every 4 weeks for up to 96 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Ipilimumab, Nivolumab, Tacrolimus, and Prednisone
Number analyzed (Participants) | 6
Participants
  Complete or Partial Response (CR or PR) | 2
  Progressive Disease (PD) | 4

7. Secondary Outcome: Rate of Allograft Loss After Receiving Ipilimumab, Nivolumab, Tacrolimus, and Prednisone
Description: Number of patients who experienced allograft loss after receiving nivolumab, ipilimumab, tacrolimus, and prednisone.
Time Frame: Up to 3 years
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab, Nivolumab, Tacrolimus, and Prednisone
Number analyzed (Participants) | 6
Participants
  Experienced allograft loss | 3
  Did not experience allograft loss | 3

ADVERSE EVENTS:
Time Frame: Up to 3 years
Groups:
- Nivolumab, Tacrolimus, and Prednisone: Patients received low-dose tacrolimus (serum trough goal 2-5 ng/mL), prednisone 5mg by mouth once a day, and nivolumab 480mg by infusion every 4 weeks for up to 96 weeks in the absence of disease progression or unacceptable toxicity.
- Ipilimumab, Nivolumab, Tacrolimus, and Prednisone: Patients received low-dose tacrolimus (serum trough goal 2-5 ng/mL), prednisone 5mg by mouth once a day, nivolumab 3 mg/kg by infusion and ipilimumab 1 mg/kg by infusion every 3 weeks for 4 doses followed by maintenance nivolumab 480mg by infusion every 4 weeks for up to 96 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Nivolumab, Tacrolimus, and Prednisone | Ipilimumab, Nivolumab, Tacrolimus, and Prednisone
All-Cause Mortality (participants affected / at risk) | 4/10 | 3/6
Serious Adverse Events (participants affected / at risk) | 6/10 | 6/6
Other Adverse Events (participants affected / at risk) | 9/10 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab, Tacrolimus, and Prednisone (N=10) | Ipilimumab, Nivolumab, Tacrolimus, and Prednisone (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac troponin (Investigations) | 0 | 1
Cardiac chest pain (Cardiac disorders) | 0 | 1
Confusion (Psychiatric disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 3 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 1
Inferior vena cava stenosis (Cardiac disorders) | 0 | 1
Lactic acidosis (Cardiac disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Pseudoaneurysm (Vascular disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 2 | 1
Skin infection (Infections and infestations) | 0 | 2
Small bowel obstruction (Gastrointestinal disorders) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Suspected allograft rejection (Renal and urinary disorders) | 1 | 2
Urinary hesitancy (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral gastroenteritis (Gastrointestinal disorders) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab, Tacrolimus, and Prednisone (N=10) | Ipilimumab, Nivolumab, Tacrolimus, and Prednisone (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 5 | 3
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bleeding at VasCath Site (Blood and lymphatic system disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood Urea Nitrogen Increased (Renal and urinary disorders) | 0 | 1
Cardiac troponin I increased (Investigations) | 3 | 2
Cheilitis (Gastrointestinal disorders) | 1 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Corneal dellan, right eye (Eye disorders) | 0 | 1
CPK increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 3 | 4
Cystitis (Renal and urinary disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Edema face (General disorders) | 0 | 2
Edema limbs (General disorders) | 1 | 2
Eye conjunctival tumor (Eye disorders) | 0 | 1
Eye redness (Eye disorders) | 0 | 1
Fatigue (General disorders) | 4 | 1
Fever (General disorders) | 3 | 1
Gait disturbance (General disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Hematuria (Renal and urinary disorders) | 1 | 2
Hepatocellular Liver Injury (Hepatobiliary disorders) | 0 | 1
Hot flashes (Vascular disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Localized edema (General disorders) | 1 | 1
Loose Stools (Gastrointestinal disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Neck stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neutrophil Count Increased (Blood and lymphatic system disorders) | 1 | 1
Pain (General disorders) | 2 | 1
Porocarcinoma (Skin and subcutaneous tissue disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 1
Thyroid stimulating hormone increased (Investigations) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumor Malodor (Skin and subcutaneous tissue disorders) | 1 | 1
Tumor Odor (General disorders) | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary hesitancy (Renal and urinary disorders) | 1 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
White Blood cell Count Increased (Blood and lymphatic system disorders) | 0 | 1
Wound infection (Infections and infestations) | 1 | 2

LIMITATIONS AND CAVEATS:
The second treatment period where participants received ipilimumab, nivolumab, tacrolimus, and prednisone was optional.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT03816332/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT03816332/ICF_001.pdf